CLINICAL TRIAL: NCT04814394
Title: The Significance of T-follicular Helper and T-follicular Regulatory Cells in Autoimmune Haemolytic Anemia
Brief Title: The Significance of Release of T-follicular Helper and T-follicular Regulatory Cells in Autoimmune Haemolytic Anemia Before and After Tratment
Acronym: fhfr
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed gamal, Doctor, Assiut University
Other Study IDs: fhraha
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Autoimmune Hemolytic Anemia
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: flowcytometry — The study of CD4,CD25,FOXP3 and PD-1 on peripheral blood sample

SUMMARY:
we study the circulating T-follicular regulatory and T-follicular regulatory cells in autoimmune hemolytic anemia.

DETAILED DESCRIPTION:
Autoimmune hemolytic anemia (AIHA) is an acquired autoimmune disease resulting in the production of antibodies directed against the patient's red blood cells (RBCs) causing shortened erythrocyte lifespan.

The main pathogensis of the disease is autoantibodies (Ab) that directed against erythrocytes, with or without complement (C) activation. The most common form of AIHA is warm AIHA characterized by the presence of warm-type autoantibodies-immunoglobulin G (IgG) which reacts optimally at 37 °C, causing RBC extravascular destruction by tissue macrophages .

Previous studies of the etiology and pathogenesis of AIHA have focused on the autoreactive B cells that have escaped tolerance mechanisms and regulatory T cells (Treg).

The main treatment of AIHA includes RBC transfusion and immune system inhibitors such as corticosteroids. During an immune response, CD4 Th cells can differentiate into several unique effector lineages that promote different immune responses via the secretion of distinct types of cytokines.

T follicular helper (Tfh) cells are a CD4 T cell lineage whose major function is to help B cells form germinal centers (GCs) and produce high-affinity antibodies(6). Tfh cells are characterized by expression of the CXCR5, the transcriptional repressor B cell lymphoma 6 (Bcl-6), programmed death 1 (PD-1), and inducible costimulator (ICOS).

Follicular regulatory T (Tfr) cells are a newly identified subset of Treg cells that coexpress markers of both Treg cells and Tfh cells. In addition to expressing Tfh-related markers, Tfr cells also express regulatory markers, such as FoxP3, CD25, CTLA-4, IL-10, and transforming growth factor β (TGFβ).

TFR cells represent a highly specialized subpopulation of Foxp3+ Tregs that co-express TFHfeatures, such as Bcl-6, CXCR5, ICOS, PD-1 and Treg features CD25 and Foxp3. TFR cells have the ability to inhibit TFH activation and cytokines production and suppress B cell GL7 and B7-1 expression and limited class switch recombination occurring in the GC via high expression of cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) and production of inhibitory cytokine- interleukin 10 (IL-10) and transforming growth factorβ (TGFβ)(5). The involvement of TFR cells in the pathogenesis of human autoimmune diseases remains speculative, but an alteration of the TFR:TFH ratio is observed in the blood of patients suffering from several autoimmune diseases, such as child immune thrombocytopenia, and rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as autoimmune hemolytic anemia, primary or secondary, male or female, any age but not on treatment

Exclusion Criteria:

* Pregnancy or breast-feeding women
* Patients treated with corticoids or immunosuppressant.
* Patients with hematological malignance.
* Patients with alloimmune hemolytic anemia as ABO incompatibility or transplant patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The sample size is 50 (25 in each arm) but number of controls will be decreased and number of cases will be increased
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of circulating T-follicular helper and T-follicular regulatory in patients with Autoimmune Hemolytic Anemia (AIHA), at diagnosis and after treatment | Baseline

SECONDARY OUTCOMES:
Measure the ratio between the T- follicular helper and T-follicular regulatory | Baseline